CLINICAL TRIAL: NCT02363569
Title: The Prognosis of Early Pregnancy With Post Coital Bleeding Compared to Early Pregnancy With Spontaneous Bleeding
Brief Title: The Prognosis of Early Pregnancy With Post Coital Bleeding
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MeirMc 180-12
Record Dates: First submitted 2015-02-02; First posted 2015-02-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2014-12

CONDITIONS: Vaginal Bleeding During Pregnancy; Postcoital Bleeding
Keywords: post coital bleeding; vaginal bleeding
MeSH Terms: conditions — Uterine Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- case-: Pregnant women (age 18-40) at 4-23 weeks of pregnancy that have appealed to the "Women ER" 24 hours after bleeding or bleeding secretions due to intercourse.
- control: Pregnant women (age 18-40) at 4-23 weeks of pregnancy that have appealed the "women ER" due to spontaneous bleeding or bleeding secretions

SUMMARY:
This is a prospective study, where the investigators will monitor pregnant women at 4-23 weeks of pregnancy coming to the "Women- E.R." at "Meir" Hospital due to spontaneous -or after intercourse- bleeding or bleeding secretions. The women will fill out questionnaires regarding past illness, vaginal bleeding, and gynecologic history. Then they will undergo full examination including ultrasound. After discharge, the investigators will recommend to all the women who came due to bleeding or bleeding secretions to avoid intercourse for two weeks after the bleeding stops. Afterwards they will be monitored until their delivery date (filling questionnaires a month after coming to the E.R. and at the end of the pregnancy). After they give birth the investigators will assess the rate of pregnancy, obstetric and embryonic complications in each of the study groups.

DETAILED DESCRIPTION:
This is a prospective study, where the investigators will monitor pregnant women at 4-23 weeks of pregnancy coming to the "Women E.R" at "Meir" Hospital due to spontaneous -or after intercourse bleeding - bleeding secretions. The women will be divided in to two groups

1. Pregnant women (age 18-40) at 4-23 weeks of pregnancy with spontaneous bleeding or bleeding secretions
2. Pregnant women (age 18-40) at 4-23 weeks of pregnancy that have appealed to the "Women ER" 24 hours after bleeding or bleeding secretions due to intercourse.

The women will fill out questionnaires regarding past illness, vaginal bleeding, and gynecologic history. Then they will undergo full examination including ultrasound. After discharge, the investigators will recommend to all the women who came due to bleeding or bleeding secretions to avoid intercourse for two weeks after the bleeding stops. Afterwards they will be monitored until their delivery date (filling questionnaires a month after coming to the E.R. and at the end of the pregnancy) The doctor that had examined the women, will have to fill out questionnaires regarding the bleeding source, the time after intercourse, how long after the intercourse the bleeding had appeared and which kind of examination he had carried out.

A month after their appeal to the E.R. and after they give birth ,the investigators will assess the rate of pregnancy, obstetric and embryonic complications in each of the study groups, by phone.

ELIGIBILITY:
Inclusion Criteria:

* women (age 18-40) with early pregnancy (4-23 weeks) with singleton or twins pregnancy that address to the "Women E.R." due to vaginal bleeding.

Exclusion Criteria:

* age >40 or <18
* women with history of more then 3 abortions.
* women with history of more then 2 pre term labor
* ectopic pregnancy
* placental previa
* women who takes anticoagulation therapy
* women with known pathology at cervix.
* women with known uterus defect. pregnancies with chromosomal defects or birth defects that was discovered at the screening tests.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with early pregnancy (4-23 weeks) with singletons or twins that address to the "Women E.R." due to vaginal bleeding.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy Complications (abortion, pre eclampsia, pre term labor,, cervix shortening, gestational diabetes, placental abruption, P-PROM(pre mature rupture of membrane), intrauterine growth retardation , Hypertension) | after they give birth (8 month after they address to the E.R.)
  abortion, pre eclampsia, pre term labor,, cervix shortening, gestational diabetes, placental abruption, P-PROM(pre mature rupture of membrane), intrauterine growth retardation , Hypertension
Delivery Complications (cesarean section,assisted delivery) | after they give birth (8 month after they address to the E.R.)
  cesarean section,assisted delivery.
Newborn Complications (low apgar, small gestational age , need for blood transfusion, artificial respiration, infection) | after they give birth (8 month after they address to the E.R.)
  low apgar, small gestational age , need for blood transfusion, artificial respiration, infection

CONTACTS AND LOCATIONS:
Overall Officials: Meir Pomeranz, M.D, Principal Investigator — Meir Hospital, Israel
Locations (1):
- Meir Hospital, Kfar Saba, Israel, Israel

REFERENCES:
- [Background] Everett C. Incidence and outcome of bleeding before the 20th week of pregnancy: prospective study from general practice. BMJ. 1997 Jul 5;315(7099):32-4. doi: 10.1136/bmj.315.7099.32. PMID 9233324
- [Background] SPEERT H, GUTTMACHER AF. Frequency and significance of bleeding in early pregnancy. J Am Med Assoc. 1954 Jun 19;155(8):712-5. doi: 10.1001/jama.1954.03690260004002. No abstract available. PMID 13162785
- [Background] Rosenthal AN, Panoskaltsis T, Smith T, Soutter WP. The frequency of significant pathology in women attending a general gynaecological service for postcoital bleeding. BJOG. 2001 Jan;108(1):103-6. doi: 10.1111/j.1471-0528.2001.00008.x. PMID 11212982